CLINICAL TRIAL: NCT05696366
Title: Combination Adjunctive Therapy to Address Multiple Metabolic Imbalances in Type 1 Diabetes
Acronym: SOTA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Lexicon Pharmaceuticals (Industry); Breakthrough T1D (Other)
Responsible Party: Principal Investigator, Schafer Boeder, Assistant Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 806355
Record Dates: First submitted 2023-01-09; First posted 2023-01-25 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; volagidemab

STUDY DESIGN:
Intervention Model Description: Each participant will receive 12-week insulin-adjunctive treatment with both: (1) SGLTi (sotagliflozin 200 mg PO each day) + Placebo and (2) SGLTi + GRA (volagidemab 35 mg subcutaneously each week), in a random-order, cross-over design with a 14-week washout period between treatment periods.
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- sotagliflozin 200 mg (Active Comparator): Each participant will receive 12-week insulin-adjunctive treatment with both: (1) SGLTi (sotagliflozin 200 mg PO each day) + Placebo and (2) SGLTi + GRA (volagidemab 35 mg subcutaneously each week), in a random-order, cross-over design with a 14-week washout period between treatment periods.
  Sotagliflozin is a dual sodium-glucose co-transporter-1 and sodium-glucose co-transporter-2 (SGLT1/2) inhibitor.
  Interventions: Drug: Sotagliflozin
- volagidemab 35 mg (Active Comparator): Each participant will receive 12-week insulin-adjunctive treatment with both: (1) SGLTi (sotagliflozin 200 mg PO each day) + Placebo and (2) SGLTi + GRA (volagidemab 35 mg subcutaneously each week), in a random-order, cross-over design with a 14-week washout period between treatment periods.
  Volagidemab is a human monoclonal antibody glucagon receptor antagonist (GRA).
  Interventions: Drug: Volagidemab
- Placebo (Placebo Comparator): Each participant will receive 12-week insulin-adjunctive treatment with both: (1) SGLTi (sotagliflozin 200 mg PO each day) + Placebo and (2) SGLTi + GRA (volagidemab 35 mg subcutaneously each week), in a random-order, cross-over design with a 14-week washout period between treatment periods.
  Interventions: Drug: Volagidemab

INTERVENTIONS:
Drug: Sotagliflozin — Sotagliflozin is a dual sodium-glucose co-transporter-1 and sodium-glucose co-transporter-2 (SGLT1/2) inhibitor.
  Arms: sotagliflozin 200 mg
Drug: Volagidemab — Volagidemab is a human monoclonal antibody glucagon receptor antagonist (GRA).
  Arms: Placebo; volagidemab 35 mg

SUMMARY:
This is a single site, double-blind, placebo-controlled, crossover trial to quantify the effects of combination adjunctive therapy on glycemic control, ketogenesis during insulinopenia, insulin resistance, and diabetes burden and quality of life.

DETAILED DESCRIPTION:
This is a single site, double-blind, placebo-controlled, crossover trial to quantify the effects of combination adjunctive therapy on glycemic control, ketogenesis during insulinopenia, insulin resistance, and diabetes burden and quality of life.

Up to 22 adult participants with type 1 diabetes (T1D) will be enrolled with at least 16 participants completing the study in full. After screening, baseline data (A1c, CGM, ambulatory insulin dosing, ambulatory ketones [fasting and after infusion set change], and psychosocial questionnaires) will be collected and participants will complete an insulin withdrawal test (IWT) and a hyperinsulinemic-euglycemic clamp (HEC) with indirect calorimetry (IDC). Participants will then receive 12-week insulin-adjunctive treatments with both: (1) SGLTi (sotagliflozin 200 mg daily) + Placebo and (2) SGLTi + GRA (volagidemab 35 mg weekly), in a random-order, cross-over design with a 14-week washout period between treatment periods. Throughout the treatment periods subjects will be seen weekly in clinic for medication dosing (GRA or placebo) and download/review of CGM, insulin, and ketone data. At the end of each treatment period, the baseline studies will be repeated. Subjects will return for a safety follow up visit 6 weeks after the final GRA or placebo dose.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 70 years old, inclusive, at the time of screening;
2. Females of non-childbearing potential must be ≥ 1 year post-menopausal or documented as being surgically sterile. Females of childbearing potential must agree to use two methods of contraception during the entire study and for an additional 3 months after the end of dosing with the investigational product;
3. Male subjects must be willing to use clinically acceptable method of contraception during the entire study and for an additional 6 months after the end of the treatment period;
4. Diagnosed with Type 1 diabetes based on clinical history or as defined by the current American Diabetes Association (ADA) criteria;
5. Treatment with a stable insulin regimen for at least 8 weeks before screening with continuous subcutaneous insulin infusion (CSII) via an insulin pump or hybrid closed loop system;
6. Currently using a Continuous Glucose Monitoring (CGM) system;
7. A1c > 7% and ≤ 10%
8. eGFR ≥ 60 mL/min/1.73m²;
9. Able to provide written informed consent approved by an Institutional Review Board (IRB).

Exclusion Criteria:

1. History or evidence of clinically significant disorder or condition that, in the opinion of the Investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion;
2. History of pancreatitis, medullary thyroid carcinoma or liver disease;
3. Clinically significant diagnosis of anemia (Hemoglobin < 9 g/dl at screening);
4. Body Mass Index (BMI) < 18.5 kg/m2 and/or weight <50kg;
5. Body Mass Index (BMI) > 35 kg/m2
6. Whole blood donation of 1 pint (500 mL) within 8 weeks prior to Screening. Donations of plasma, packed RBCs, platelets or quantities less than 500 mL are allowed at investigator discretion;
7. Current or recent (within 1 month of screening) use of diabetes medications other than insulin; (examples include GLP-1 RA, SGLT-2i, Pramlintide, Metformin);
8. Women who are pregnant or lactating/breastfeeding;
9. Unable or unwilling to follow the study protocol or who are non-compliant with screening appointments or study visits;
10. Any other condition(s) that might reduce the chance of obtaining study data, or that might cause safety concerns, or that might compromise the ability to give truly informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 12 weeks
  Quantify the effects of combination adjunctive therapy on glycemic control. Though it has limitations, the HbA1c remains the gold standard measurement of glycemic control in diabetes.

SECONDARY OUTCOMES:
Change in percent time in range (70-180 mg/dl) by CGM | 12 weeks
  Continuous glucose monitoring (CGM) provides much more granular data relating to glucose trends and time spent in target glucose range, above range (hyperglycemia), and below range (hypoglycemia).
Change in subject self reported ambulatory insulin dosing | 12 weeks
  Change in ambulatory insulin dosing as shown through subject insulin diary.

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Altman Clinical & Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
Will not share IPD